CLINICAL TRIAL: NCT04873778
Title: Comparing Effects of Kinesio and Dynamic Tapings in Postpartum Women With Pelvic Girdle Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, YI-JU TSAI, associate professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCKU-Taping
Record Dates: First submitted 2021-04-27; First posted 2021-05-05 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Pelvic Girdle Pain
Keywords: Kinesio taping; Dynamic taping; Postpartum
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dynamic taping group (Experimental): stabilize the Sacroiliac joints and stimulate muscle contraction
  Interventions: Device: Dynamic taping
- kinesio taping group (Experimental): stabilize the Sacroiliac joints and stimulate muscle contraction
  Interventions: Device: Kinesio taping
- control group (Placebo Comparator): use Kinesio taping for placebo effect
  Interventions: Device: Kinesio taping

INTERVENTIONS:
Device: Kinesio taping — Kinesio taping: Invented by Japan Dr.Kase, increase circulation by creating lifts skin,release pain and inflammation, stabilize joints
  Arms: control group; kinesio taping group
Device: Dynamic taping — Dynamic taping: Invented by Kendrick,elasticised with multi-directional rebound and with strong elastic resistance and recoil than KT
  Arms: Dynamic taping group

SUMMARY:
About 45% of pregnant women and 25% of women postpartum suffer from Pelvic girdle pain. Pain is often reported to be localized between costal margin and gluteal fold with or without radiation to lower limb or symphysis pubic. Kinesio taping (KT) is the application of an elastic tape, for treating musculoskeletal conditions through enhancing muscle strength, relieving spasms, pain and edema, improving blood circulation and lymph reflux, as well as stabilizing joints. However, with limited evidence and a lack of well-designed study, the effects of KT in postpartum women with PGP remains unclear. Compared with KT, the dynamic taping(DT) is recently developed and has stronger elastic resistance and recoil. The DT may have better effects than the KT, although this notion has not been examined. In this study, we make a hypothesis that PGP women in the DT group would have better improvements on pain, disability, quality of life, and PFM functions than that in the KT group and control group.

DETAILED DESCRIPTION:
The main purpose for this study are to investigate the effects of KT and DT on pain, disability, physical functions, and quality of life, as well as PFM functions in postpartum women with PGP. 60 postpartum women with PGP will be randomized into one of the three groups:(1) kinesio taping group,(2) dynamic taping group (3)control group, and receive 4 weeks intervention. All participants will receive 3 assessments at the baseline, immediately after first taping session, and after 4-week interventions. The outcome measures will include Visual Analog Scale measures of pain intensity, Pelvic Girdle Questionnaire/ Oswestry Disability Index/ Patient specific functional scale measures and Global rating of change score. for disability. The quality of life will be measured by 36-item Short-Form Survey， The Physical functions include Active Straight Leg Raise Fatigue task , Time up and go test,10-meter walk test. The PFM functions will be measured by Modified Oxford grading scale and Perineometer. It is expected that PGP women in both the KT group and DT group will have more improvements than the control group. But the DT group will have even more improvements than the KT groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age: > 20 year
2. Postpartum:≥ 3 months
3. Pain onset during pregnancy
4. Pain location is located between costal margin and gluteal fold with or without radiation to lower limb or symphysis pubic
5. Clinical screening test for pelvic pain :

Active Straight Leg Raising : positive

* 2 (+) posterior pelvic pain provocation tests (+ symphysis ≥ 1)

Exclusion Criteria:

1. BMI ≥ 30
2. lumbar or pelvic surgery
3. History of fracture
4. Radiculopathy or myopathy
5. Gynaecological disorders
6. Serious cardiovascular disease
7. Tumors
8. Diagnosed psychiatric disease
9. Ongoing pregnancy
10. Allergy to acrylic

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Change from baseline pain intensity up to 4 weeks
  for pain
Pelvic Girdle Questionnaire | Change from disability baseline up to 4 weeks
  for disability
Oswestry Disability Index | Change from baseline disability up to 4 weeks
  for disability
Patient specific functional scale measures | Change from baseline disability up to 4 weeks
  for disability
Global rating of change score | Change from baseline disability up to 4 weeks
  for disability
36-item Short-Form Survey | Change from baseline quality of life up to 4 weeks
  for quality of life
Active Straight Leg Raise Fatigue task | Change from baseline Physical functions up to 4 weeks
  for Physical functions
Time up and go test | Change from baseline Physical functions up to 4 weeks
  for Physical functions
10-meter walk test | Change from baseline Physical functions up to 4 weeks
  for Physical functions
Modified Oxford grading scale | Change from baseline PFM functions up to 4 weeks
  for PFM functions
Perineometer | Change from baseline PFM functions up to 4 weeks
  for PFM functions

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan